CLINICAL TRIAL: NCT05680896
Title: The Risk of SARS-CoV-2 Infection and Severity of COVID-19 Among Healthcare Workers With or Without Previous COVID-19 Vaccines
Brief Title: SARS-CoV-2 Infection Among Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Chao Wu, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 20222-746
Record Dates: First submitted 2022-12-22; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: inactivated COVID-19 vaccines; orally aerosolized Ad5-nCoV — the protection of COVID-19 vaccines on breakthrough infection

SUMMARY:
At present, COVID-19 vaccine is considered as the safest, economic and effective measure to prevent and control COVID-19. Adaptive immunity, including humoral immunity and cellular immunity, plays a role in anti-viral responses. Cellular immunity includes virus specific B cells and T cells, which can provide long-term memory immunity. For acute viral infection, neutralizing antibody is of great significance in preventing infection, while memory cell immunity can maintain a good broad-spectrum and persistence in controlling mutant strains, which is a key factor in controlling viral replication after infection and reducing severe disease and death. However, there is no systematic study on the specific immune response and infection risk of novel coronavirus, and there is no definite conclusion on which specific protective immune response induced by vaccine can reduce the risk of infection. Therefore, this study aims to establish a prospective real-world cohort, analyze the correlation between multiple baseline immune protection indicators and infection risk, follow up the population with breakthrough infection, and monitor the dynamic specific immune response to COVID-19 in peripheral blood and respiratory mucosa. This study will provide an important scientific basis for us to scientifically assess the risk of individual infection with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. SARS-CoV-2 nucleic acid testing showed negative within 72 hours

Exclusion Criteria:

1.Do not consent to enroll in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers in Nanjing Drum Tower Hospital, Nanjing, China
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-03-21 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | from Dec 2022 to April 2023
  SARS-CoV-2 infection confirmed by either by nucleic acid testing or antigen testing
The severity of COVID-19 | from Dec 2022 to April 2023
  the severity of COVID-19 symptoms including the period from SARS-CoV-2 positive to negative, fever days, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Wu, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Y, Zhao T, Chen L, Jiang G, Geng Y, Li W, Yin S, Tong X, Tao Y, Ni J, Lu Q, Ning M, Wu C. SARS-CoV-2 Omicron infection augments the magnitude and durability of systemic and mucosal immunity in triple-dose CoronaVac recipients. mBio. 2024 Apr 10;15(4):e0240723. doi: 10.1128/mbio.02407-23. Epub 2024 Mar 8. PMID 38456703